CLINICAL TRIAL: NCT05703698
Title: EEG Outcomes From Cognitive Behavioural Therapy for Psychosis
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ontario Shores Centre for Mental Health Sciences (Other)
Responsible Party: Principal Investigator, Michael Best, Assistant Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38831
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-07

CONDITIONS: Psychotic Disorders; Schizophrenia and Related Disorders
Keywords: Psychosis; Electroencephalogram; CBTp; CBT
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Formulation-based CBTp will be delivered with a maximum of 30 sessions over 6 months based on an established manual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive Behavioural Therapy for psychosis (Experimental): CBTp will be delivered according to an established manual that the PI has previously used successfully for in-person treatment. Treatment will consist of individual sessions with a psychologist employed by the University of Toronto for 1-hour per week for 6-months, or by one of the listed clinical graduate students under his supervision. All treatment will be delivered in-person. This treatment will be delivered in addition to usual care and no changes to usual care will be required.
  Interventions: Behavioral: Cognitive Behavioural Therapy for Psychosis

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for Psychosis — CBT will be delivered according to an established manual that the PI has previously used successfully for in-person treatment. Treatment will consist of individual sessions with a psychologist employed by the University of Toronto for 1-hour per week for 6-months, or by one of the listed clinical graduate students under his supervision. All treatment will be delivered in-person. This treatment will be delivered in addition to usual care and no changes to usual care will be required.
  Other Names: CBT; CBTp

SUMMARY:
Despite overwhelming evidence for neurocognitive and neurophysiological factors involved in the etiology of psychosis, these factors have never been examined as mechanisms of improvement from CBTp. The first aim in the present study is to examine neurophysiological outcomes from CBTp using electroencephalography (EEG). The second aim is to examine neurocognitive outcomes from CBTp. This is an open-label pilot study. Twenty participants will receive CBTp and will be assessed at baseline and after 4 months.

DETAILED DESCRIPTION:
Despite decades of refining traditional treatments for schizophrenia-spectrum disorders, recovery rates remain unchanged at only 13.5%, and there is an urgent need for innovative new interventions. Cognitive behavioural therapy has more recently been applied to treating psychosis and initial evidence has suggested that cognitive behavioural therapy for psychosis (CBTp) is the most effective psychosocial intervention available for psychosis. However, the efficacy of CBTp has been limited to moderate effect sizes. Little is currently understood about the mechanisms of CBTp, and a greater understanding of mechanisms is necessary in order to improve treatment efficacy. Despite overwhelming evidence for neurocognitive and neurophysiological factors involved in the etiology of psychosis, these factors have never been examined as mechanisms of improvement from CBTp. Cognitive behavioural therapy for psychosis (CBTp) has demonstrated efficacy for reducing positive symptoms, negative symptoms, and improving community functioning6 for individuals diagnosed with psychotic disorders. Despite meta-analytic evidence for the efficacy of CBTp, little is known about the neurophysiological processes through which symptomatic and functional change occurs. Electroencephalography (EEG) provides temporally precise measurement of neurophysiological activity. Positive symptoms have been associated with reduced integration of discrepant information as indexed by the N400 event-related potential, reduced resting state power in the EEG alpha frequency band, and reduced cognitive control as indexed by EEG alpha and theta power during cognitive flanker tasks. Additionally, neurocognitive abilities such as attention, memory, and problem solving are the best predictors of community functioning among individuals diagnosed with psychotic disorders. Although CBTp improves community functioning,[6] neurophysiological and neurocognitive outcomes have never been examined as therapeutic mechanisms from CBTp, despite the fact that therapeutic processes would be expected to improve cognitive functions.

Aim 1: Examine neurophysiological outcomes from CBTp using EEG.

Aim 2: Examine neurocognitive outcomes from CBTp

Hypothesis 1: After CBTp it is expected that participants will have a) increased N400 amplitude; b) increased resting state EEG alpha power; and c) reduced alpha and increased theta power during a flanker task

Hypothesis 2: After CBTp participants will have increased global neurocognitive abilities as indexed by a neurocognitive composite score.

Although CBTp has demonstrated efficacy to improve symptoms for individuals experiencing psychosis, little is known about the neurophysiological process through which this improvement occurs, and neither EEG nor neurocognitive outcomes from CBTp have ever been examined. The current results will provide preliminary evidence for neurophysiological mechanisms of change from CBTp that will increase understanding of the disorder and provide critical insights for refining psychotherapeutic interventions. Additionally, psychotherapy trials typically only examine psychological outcomes, however, if CBTp is effective it would be expected that this could be detected at both the neurophysiological level and neurocognitive level as well. My incorporation of multiple levels of assessment in clinical trials was recently praised as a goldstandard approach to trial methodology. This line of research is critical to improving the efficacy of CBTp.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria is anyone who meets the criteria of schizophrenia, schizoaffective disorder or any other psychotic disorder, are also 18-65 years of age, are not abusing drugs or alcohol and can read and speak English. Participants must be experiencing active symptoms of psychosis as indicated on the PANSS.

Exclusion Criteria:

* Exclusion criteria include anyone with a neurological disease or neurological damage, medical illnesses that can change neurocognitive function, a medical history of head injury with loss of consciousness and those with physical handicaps that would prevent them from engaging in assessment procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) Total Score | Change from Baseline to Follow-up (6 months post treatment)
  The PANSS is a 30-item semi-structured interview assessing positive, negative symptoms and general psychopathology. Each item is scored on a 7-point scale (1 = absent, 2 = minimal, 3 = mild, 4 = moderate, 5 = moderate severe, 6 = severe, 7 = extreme). The lowest score would be a 30 and the highest score would be 210. A higher score would indicate increased symptomology.

SECONDARY OUTCOMES:
Personal and Social Performance Scale (PSP) | Change from Baseline to Follow-up (6 months post treatment)
  The PSP assesses community functioning through a brief interview with the participant about their daily activities. It contains 4 areas: (1) socially useful activities; including work and study; (2) personal and social relationships; (3) self-care; (4) disturbing and aggressive behaviors. The total score ranges from 1 to 100 and is interpreted on a 10-point intervals. Lower scores indicates more severe functional impairment while higher scores indicate better functioning.
The Psychotic Symptom Rating Scales (PSYRATS) | Change from Baseline to Follow-up (6 months post treatment)
  The PSYRATS assesses frequency and distress associated with the experiences of auditory hallucinations and delusions based on the PANSS interview. Each of the 17 items is scored on a 5-point scale, where a score of 0 indicates no presence, and 4 indicates the highest severity. The lowest score would be a 0 and the highest score would be 68. A higher score would indicate increased symptomology.
Calgary Depression Scale for Schizophrenia (CDSS) | Change from Baseline to Follow-up (6 months post treatment)
  The CDSS is a 9-item interview-based measure of depression symptoms specifically designed for use with people experiencing schizophrenia. Each item is scored on a 4-point scale (0 = absent, 1 = mild, 2 = moderate, 4 = severe). The lowest score would be a 0 and the highest score would be 36. A higher score would indicate increased severity of depressive symptoms.
The Questionnaire About the Process of Recovery (QPR) | Change from Baseline to Follow-up (6 months post treatment)
  QPR is a self-report measure assessing recovery with people experiencing psychosis. This version contains 22 items while the response to each statement is scored on a 5-point Likert scale ranging from "0 = strongly disagree" to "4 = strongly agree". The lowest possible score is 0 and the highest score could be 88. Higher scores would indicate better recovery.
Beliefs About Paranoia Scale (BAPS) | Change from Baseline to Follow-up (6 months post treatment)
  The BAPS is a 31-item self-report measure assessing metacognitive beliefs about paranoia. The degree of agreement to each statement is scored on a 4-point scale (1 = not at all, 2 = somewhat, 3 = moderately so, 4 = very much). Scales include positive, negative and normalizing beliefs about paranoia, and paranoia as a survival strategy. The lowest score would be 31 and the highest score would be 124. Higher scores are indicative of more beliefs and are shown to be related to paranoid ideation.
Beliefs About Voices Questionnaire (BAVQ) | Change from Baseline to Follow-up (6 months post treatment)
  BAVQ-R is a 35-item self-report measure assessing metacognitive perception, feelings about and reaction to auditory hallucinations. The degree of agreement to each statement is scored on a 4-point scale, ranging from disagree to strongly agree. Five subscales (malevolence, benevolence, omnipotence, resistance, engagement) are included. The lowest possible score is 0 and the highest score would be 105. Higher scores would indicate a tighter relationship with voices.
Experiences Questionnaire (EQ) | Change from Baseline to Follow-up (6 months post treatment)
  The EQ is a 11-item self-report measure assessing observations of thoughts and self. Frequency of experiences is scored on a 5-point scale, ranging from "1 = never" to "5 = all the time". The lowest possible score is 11 while the highest score would be 55. Higher scores would indicate increased levels of self-acceptance and mindfulness.
Brief Core Schema Scale (BCSS) | Change from Baseline to Follow-up (6 months post treatment)
  The BCSS is a 24-item self-report measure assessing positive and negative judgments individuals hold about themselves and others. Responses are first given dichotomously as "no" or "yes". "No" is scored as 0 and if the answers are "yes", the intensity of beliefs are then rated on a 4-point scale (1 = believe it slightly, 2 = believe it moderately, 3 = believe it very much, 4 = believe it totally). The lowest score would be a 0 and the highest score would be a 96. Higher scores in the positive-self subscale indicate more positive beliefs about selves, while higher scores in the negative-self subscale indicate more negative beliefs about selves. Higher scores in the positive-others subscale indicate more positive beliefs about others, while higher scores in the negative-others subscale indicate more negative beliefs about others.
Dysfunctional Attitude Scale (DAS) | Change from Baseline to Follow-up (6 months post treatment)
  DAS is a 40-item self-report measure assessing dysfunctional beliefs. The degree of agreement to each statement is scored on a 7-point Likert scale (1 = agree totally, 2 = agree very much, 3 = agree slightly, 4 = neutral, 5 = disagree slightly, 6 = disagree very much, 7 = disagree totally). The lowest possible scale is 40 while the highest possible scale is 280. Higher scores would indicate more negative beliefs.
Davos Assessment of Cognitive Biases Scale (DACOBS) | Change from Baseline to Follow-up (6 months post treatment)
  DACOBS is a 42-item self-report inventory assessing cognitive processing biases associated with psychosis. The degree of agreement to each statement is scored on a 7-point Likert scale, ranging from "1 = strongly disagree" to "7 = strongly agree". The lowest score would be a 42 and the highest score would be a 294. Higher scores would indicate more cognitive biases.
Childhood Trauma Questionnaire (CTQ) | Change from Baseline to Follow-up (6 months post treatment)
  The CTQ is a 28-item self-report measure assessing experiences of trauma during childhood. Frequency of experiences is reported on a 5-point scale, ranging from "never true" to "very often true". Reverse-coded items are included. The lowest score would be a 28 and the highest score would be a 140. Higher scores would indicate more trauma exposure.
Working Alliance Inventory (WAI) | Change from Baseline to Follow-up (6 months post treatment)
  The WAI assesses the quality of the therapeutic relationship. 36 items are to be completed both by the therapist and the client. Frequency of experiences are rated on a 7-point Likert scale (1 = never, 2 = rarely, 3 = occasionally, 4 = sometimes, 5 = often, 6 = very often, 7 = always). Reverse-coded items are included. The lowest score would be a 36 and the highest score would be a 252. Highest scores would indicate more therapeutic alliance.
Psychological Distance Scaling Task (PDST) | Change from Baseline to Follow-up (6 months post treatment)
  The PDST is an experimental task associated with cognitive processing biases in psychosis. It gives measure of both how positive and negative a person views themselves, and how tightly held these beliefs are based on the clustering of the ratings. Participants would place adjectives on the grid based on self-descriptiveness and valence, while responses ranging from "not at all like me" to "very much like me" and "very negative" to "very positive". Smaller interstimulus distances among negative self-relevant adjectives and greater interstimulus distances among positive self-relevant adjectives would indicate more negative biases about selves.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Best, Ph.D., Principal Investigator — University of Toronto
Locations (1):
- University of Toronto Scarborough, Scarborough Village, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaaskelainen E, Juola P, Hirvonen N, McGrath JJ, Saha S, Isohanni M, Veijola J, Miettunen J. A systematic review and meta-analysis of recovery in schizophrenia. Schizophr Bull. 2013 Nov;39(6):1296-306. doi: 10.1093/schbul/sbs130. Epub 2012 Nov 20. PMID 23172003
- [Background] Alvarez-Jimenez M, Parker AG, Hetrick SE, McGorry PD, Gleeson JF. Preventing the second episode: a systematic review and meta-analysis of psychosocial and pharmacological trials in first-episode psychosis. Schizophr Bull. 2011 May;37(3):619-30. doi: 10.1093/schbul/sbp129. Epub 2009 Nov 9. PMID 19900962
- [Background] van der Gaag M, Valmaggia LR, Smit F. The effects of individually tailored formulation-based cognitive behavioural therapy in auditory hallucinations and delusions: a meta-analysis. Schizophr Res. 2014 Jun;156(1):30-7. doi: 10.1016/j.schres.2014.03.016. Epub 2014 Apr 14. PMID 24731619
- [Background] Morrison AP, Turkington D, Pyle M, Spencer H, Brabban A, Dunn G, Christodoulides T, Dudley R, Chapman N, Callcott P, Grace T, Lumley V, Drage L, Tully S, Irving K, Cummings A, Byrne R, Davies LM, Hutton P. Cognitive therapy for people with schizophrenia spectrum disorders not taking antipsychotic drugs: a single-blind randomised controlled trial. Lancet. 2014 Apr 19;383(9926):1395-403. doi: 10.1016/S0140-6736(13)62246-1. Epub 2014 Feb 6. PMID 24508320
- [Background] Grant PM, Huh GA, Perivoliotis D, Stolar NM, Beck AT. Randomized trial to evaluate the efficacy of cognitive therapy for low-functioning patients with schizophrenia. Arch Gen Psychiatry. 2012 Feb;69(2):121-7. doi: 10.1001/archgenpsychiatry.2011.129. Epub 2011 Oct 3. PMID 21969420
- [Background] Morrison AP, Law H, Carter L, Sellers R, Emsley R, Pyle M, French P, Shiers D, Yung AR, Murphy EK, Holden N, Steele A, Bowe SE, Palmier-Claus J, Brooks V, Byrne R, Davies L, Haddad PM. Antipsychotic drugs versus cognitive behavioural therapy versus a combination of both in people with psychosis: a randomised controlled pilot and feasibility study. Lancet Psychiatry. 2018 May;5(5):411-423. doi: 10.1016/S2215-0366(18)30096-8. Epub 2018 Apr 5. PMID 29605187
- [Background] Jackson F, Foti D, Kotov R, Perlman G, Mathalon DH, Proudfit GH. An incongruent reality: the N400 in relation to psychosis and recovery. Schizophr Res. 2014 Dec;160(1-3):208-15. doi: 10.1016/j.schres.2014.09.039. Epub 2014 Oct 22. PMID 25449716
- [Background] Bowie CR, Reichenberg A, Patterson TL, Heaton RK, Harvey PD. Determinants of real-world functional performance in schizophrenia subjects: correlations with cognition, functional capacity, and symptoms. Am J Psychiatry. 2006 Mar;163(3):418-25. doi: 10.1176/appi.ajp.163.3.418. PMID 16513862
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Nuechterlein KH, Green MF, Kern RS, Baade LE, Barch DM, Cohen JD, Essock S, Fenton WS, Frese FJ 3rd, Gold JM, Goldberg T, Heaton RK, Keefe RS, Kraemer H, Mesholam-Gately R, Seidman LJ, Stover E, Weinberger DR, Young AS, Zalcman S, Marder SR. The MATRICS Consensus Cognitive Battery, part 1: test selection, reliability, and validity. Am J Psychiatry. 2008 Feb;165(2):203-13. doi: 10.1176/appi.ajp.2007.07010042. Epub 2008 Jan 2. PMID 18172019
- [Background] Vinogradov S. Has the Time Come for Cognitive Remediation in Schizophrenia...Again? Am J Psychiatry. 2019 Apr 1;176(4):262-264. doi: 10.1176/appi.ajp.2019.19020160. No abstract available. PMID 30929502
- [Background] Kim M, Lee TY, Lee S, Kim SN, Kwon JS. Auditory P300 as a predictor of short-term prognosis in subjects at clinical high risk for psychosis. Schizophr Res. 2015 Jul;165(2-3):138-44. doi: 10.1016/j.schres.2015.04.033. Epub 2015 May 5. PMID 25956629
- [Background] Scherbaum S, Fischer R, Dshemuchadse M, Goschke T. The dynamics of cognitive control: evidence for within-trial conflict adaptation from frequency-tagged EEG. Psychophysiology. 2011 May;48(5):591-600. doi: 10.1111/j.1469-8986.2010.01137.x. Epub 2010 Nov 2. PMID 21044093
- [Background] Morrison AP, French P, Walford L, Lewis SW, Kilcommons A, Green J, Parker S, Bentall RP. Cognitive therapy for the prevention of psychosis in people at ultra-high risk: randomised controlled trial. Br J Psychiatry. 2004 Oct;185:291-7. doi: 10.1192/bjp.185.4.291. PMID 15458988
- [Background] Blackburn, I., James, I., Milne, D., Baker, C., Standart, S., Garland, A., & Reichelt, F. The revised cognitive therapy scale (CTS-R): Psychometric properties. Behavioural and Cognitive Psychotherapy. 2001; 29(4): 431-446.